CLINICAL TRIAL: NCT00624715
Title: Cannabinoid Receptor Function & Alcoholism: Effects of Δ-9-THC
Brief Title: Cannabinoid Receptor Function & Alcoholism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0707002888
Record Dates: First submitted 2008-02-18; First posted 2008-02-27 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- THC (Active Comparator): * High dose: 0.036 mg/kg (2.5 mg in a 70 kg individual) IV (in the vein) dissolved in ethanol.Equivalent to smoking a full joint
  * Low dose: 0.018 mg/kg (1.25 mg in a 70kg individual)IV (in the vein) dissolved in ethanol.Equivalent to smoking ½ of a joint
  * Very low dose: 0.0036 mg/kg (0.25 mg in a 70 kg individual)IV (in the vein) dissolved in ethanol.Equivalent to smoking 1/10 of a joint
  Interventions: Drug: THC
- Placebo (Placebo Comparator): Placebo: Small amount of ethanol IV (in the vein), (quarter teaspoon).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC — * High dose: 0.036 mg/kg (2.5 mg in a 70 kg individual)IV (in the vein) dissolved in ethanol. Equivalent to smoking a full joint
  * Low dose: 0.018 mg/kg (1.25 mg in a 70kg individual) IV (in the vein) dissolved in ethanol.Equivalent to smoking ½ of a joint
  * Very low dose: 0.0036 mg/kg (0.25 mg in a 70 kg individual)IV (in the vein) dissolved in ethanol. Equivalent to smoking 1/10 of a joint
  Arms: THC
Drug: Placebo — Placebo: Small amount of ethanol IV (in the vein), (quarter teaspoon).
  Arms: Placebo

SUMMARY:
This study attempts to characterize the effects of tetrahydrocannabinol (THC). Tetrahydrocannabinol is the active ingredient of marijuana, cannabis, "ganja", or "pot". This study will involve healthy volunteers who 1) have no history of alcoholism in their family or 2) have a family history of alcoholism. This study looks at individuals with or without a family history of alcoholism to determine if there is a difference between the two groups in the response to THC.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to cannabis at least once

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2007-08-09 (Actual); Primary Completion 2010-06-22 (Actual); Study Completion 2010-06-22 (Actual)

PRIMARY OUTCOMES:
Clinician Administered Dissociative Symptoms Scale, Visual Analog Scale ("High" rating), Rey Auditory Verbal Learning Test | Baseline, +15, +25 (RAVLT only), +70, +240

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States